CLINICAL TRIAL: NCT00663364
Title: Klinische Untersuchung Zur Pflege Trockener Haut Mit Physiogel AI Lotion Und Physiogel Lotion
Brief Title: Care of the Dry Skin With Physiogel AI Lotion® (W0156)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sonja Ständer, Prof. Dr., Department of Dermatology, University of Münster
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SST-Pr-5-2006
Record Dates: First submitted 2008-04-14; First posted 2008-04-22 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2009-02

CONDITIONS: Eczema
Keywords: dry skin
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): Physiogel AI Lotion
  Interventions: Drug: Physiogel AI Lotion, Physiogel Lotion
- II (Active Comparator): Physiogel Lotion twice daily
  Interventions: Drug: Physiogel AI Lotion, Physiogel Lotion

INTERVENTIONS:
Drug: Physiogel AI Lotion, Physiogel Lotion — Physiogel AI Lotion and Physiogel Lotion is a cosmetic, applied twice daily to dry skin

SUMMARY:
Dry skin is a physiological condition and is characterized in contrast to greasy skin by roughness, desquamation and lack of brightness of the skin surface. Subjectively, feelings of tension, burning and itching can occur. Dry skin needs special care due to its structural and functional characteristics.We monitor an application test the Dermatocosmetics Oilatum Physiogel AI Lotion and Physiogel Lotion. This is to be accomplished with patients having dry skin. The influence on the roughness of skin, desquamation, feeling of tingle, burning and itching should be documented. If sleep quality is disturbed by tingle or itch, this will be monitored, too.

DETAILED DESCRIPTION:
The included patients use the lotion twice daily for a two-week period. If not sufficient it can be continued up to a four-weeks period. Additionally, the patient receives a documentation sheets to note several parameters. In a sensory assessment, product specific parameter such as spreadability, permeability, lubricating, smell of lotion and cosmetic acceptance during the treatment will be assessed (at the beginning, after 2 weeks, after 4 weeks, 2 weeks after stopping treatment). After four weeks the skin care measurement will be terminated and the patient can continue with a treatment of his choice. A monitoring of at least 50 patients per preparation is intended.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age: over 18 years
2. Willing to apply skin care for 2 to 4 weeks, twice daily
3. Willing to fulfill questionnaires / home diaries: self-perception of roughness of the skin, desquamation of the skin, lack of skin brightness, feelings of tension and itching

Exclusion Criteria:

1. Participation in any other research study during the previous 4 weeks.
2. Previous participation in this study.
3. Concurrent participation in any other research study involving an investigational product.
4. Current need for the use of topical steroids.
5. History of skin disease or allergy likely to interfere with the study or known sensitivity to the test product or its ingredients.
6. Subjects considered unable or unlikely to fulfill diaries.
7. Employees of (CRO) or Stiefel Laboratories, or an immediate family member (partner, offspring, parents, siblings or sibling's offspring) of an employee.
8. History of cancer.
9. Recent immunization (less than 10 days prior to the use of the test product).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-04; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Improvement of dry skin Improvement of burning, stinging and pruritus (if present) Improvement of quality of life | two weeks
Improvement of burning, stinging and pruritus (if present) | two weeks
Improvement of quality of life | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Ständer, MD, Principal Investigator — Department of Dermatology, University Hopsital Münster
Locations (1):
- Department of Dermatology, Münster, North Rhine-Westphalia, Germany